CLINICAL TRIAL: NCT01340196
Title: Effect of Multiple Dosing With 240 mg BID BI 201335 on the Steady State Pharmacokinetics of 300mg QD Tenofovir and Effect of Multiple Dosing With 300mg QD Tenofovir on Steady State BI 201335 Pharmacokinetics in Healthy Male and Female Volunteers
Brief Title: Drug Drug Interaction of BI 201335 and Tenofovir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1220.50
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Results first posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

ARMS (1):
- sequence 1 (Experimental): tenofovir medium dose once daily (qd) for first 15 days; BI 201335 medium dose twice daily (bid) on days 8 through day 22 (morning dose on day 22 only)
  Interventions: Drug: tenofovir/BI 201335

INTERVENTIONS:
Drug: tenofovir/BI 201335 — tenofovir medium dose once daily (qd) for first 15 days; BI 201335 medium dose twice daily (bid) on days 8 through 22 with last dose on morning of day 22

SUMMARY:
The objective of this study is to evaluate the drug-drug interaction potential between BI 201335 and concomitantly administered tenofovir which is used in treatment regimens for HIV infection and/or Hepatitis B infection. Results of this study will serve as a basis for guidance of dose adjustments or other precautionary measures when BI201335 and tenofovir are coadministered.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males and female subjects and according to medical history, including the physical examination, vital signs (blood pressure, pulse rate), 12-lead electrocardiogram and clinical laboratory tests; all with acceptable findings.
2. Age =18 to =55 years
3. Weighing at least 50 kg, and body mass index >=18.5 and BMI <=29.9 kg/m2 (Body Mass Index).
4. Volunteers must not leave the research unit, during the entire length of the study and must be willing to comply with the protocol and complete all study-related activities.

Exclusion criteria:

1. Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram) deviating from normal and of clinical relevance, as assessed by the investigator.
2. Active diseases of the gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, musculoskeletal, immunologic, rheumatologic, hormonal, neurological system, clinically relevant electrolyte disorders or bleeding disorders that require current medical treatment.
3. Diseases of the central nervous system or psychiatric disorders.
4. History of photosensitivity or recurrent rash.
5. History of orthostatic hypotension, fainting spells or blackouts.
6. Chronic or clinically relevant acute infections.
7. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant.
8. Intake of drugs with a long half-life >24:00 hours within at least one month or less than ten half lives of the respective drug before enrollment in the study (with the exception of hormonal contraceptives).
9. Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment as nutraceuticals and herbal remedies that would interfere with either the absorption, distribution or metabolism of BI 201335 NA, or that prolong the QT/QTc interval.
10. Use of any investigational drug within 30 days prior to enrollment; or the planned use of any investigational drug during the course of the current study.
11. Smoking (>10 cigarettes or >3 cigars or >3 pipes/day)
12. Inability to abstain from smoking more than 3 cigarettes/day during the period of dosing with study medication.
13. Drug and alcohol abuse (>60g/day).
14. Blood donation (more than 100 mL within four weeks prior to administration or during the trial).
15. Excessive physical activities within one week prior to administration or during the trial.
16. Any laboratory value outside the reference range that is of clinical relevance at screening, according to the judgment of the investigator, and in consultation with the clinical monitor.
17. Known elevated liver enzymes in past with any compound (experimental or marketed).
18. Concomitant administration of any food product known to alter P450 enzyme activity such as grapefruit juice, Seville oranges, St. John's Wort.
19. Concomitant administration of oral contraceptives (subjects who stopped oral contraceptives at least 7 days prior to Day 1 may be included.
20. Inadequate venous access.
21. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTcF, or QTcB interval >450 ms).
22. Infection with hepatitis B (HBV), or hepatitis C virus (HCV),
23. Positive test for HIV-1 or HIV-2. For women of child bearing potential (WOCBP)
24. Pregnancy or planning to become pregnant within 2 months of study completion
25. Positive pregnancy test at screening visit
26. No proof of sterilization, or not willing or unable to consistently use an acceptable method of double barrier contraception including IUD, or diaphragm with spermicidal cream/jelly and condoms for male partner, during and up to 3 months after completion/termination of the trial.
27. Lactation period with active breastfeeding from time of screening to 30 days after end of trial visit.

    For male subjects
28. No proof of sterilization, or not willing or unable to consistently use an acceptable method of double barrier contraception including a condom each time and female partner of child bearing potential consistently uses oral birth control pills, or an IUD, or a diaphragm with spermicidal cream/jelly). Male subjects must not father a child from administration of the first dose and up to 3 months after the last dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1220.50.0001 Boehringer Ingelheim Investigational Site, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: tenofovir medium dose (300mg) once daily (qd, oral) for first 15 days; Faldaprevir starting dose of 480mg and evening dose of 240mg on day 8; medium dose (300mg) twice daily (bid) on days 9 through day 22 (morning dose on day 22 only)
Period: Treat. Period 1 (Tenofovir)
Arm/Group | All Participants
Started | 16
Completed | 16
Not Completed | 0
Period: Treat. Period 2 (Tenofovir/Faldaprevir)
Arm/Group | All Participants
Started | 16
Completed | 16
Not Completed | 0
Period: Treat. Period 3 (Faldaprevir)
Arm/Group | All Participants
Started | 16
Completed | 14
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Steady-state Pharmacokinetics of AUC0-24 of Tenofovir on Day 7 and on Day 15
Description: Area under the concentration-time curve (AUC) of the analyte in plasma over the time interval 0-24 hours, at steady state.
Time Frame: 144:00, 144:30, 145:00, 145:30, 146:00, 147:00, 148:00, 150:00, 152:00, 156:00, 168:00 hours on day 7 and 168:00, 168:30, 169:00, 169:30, 170:00, 172:00, 174:00, 176:00, 178:00, 180:00, 192:00 hours on day 15
Population: All participants from the pharmacokinetic analysis set (PK set), including all subjects who were documented to have taken at least one dose of trial medication (treated set) who provided evaluable data for at least 1 observation for at least 1 primary PK endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Tenofovir: tenofovir medium dose (300mg) once daily (qd) (day 1 to 7)
- Tenofovir/Faldaprevir: tenofovir medium dose (300mg) once daily (qd) (day 8 to 15); Faldaprevir starting dose of 480mg and evening dose of 240mg on day 8; medium dose (240mg) twice daily (bid) on days 9 through day 15
- Faldaprevir: Faldaprevir medium dose (240mg) twice daily (bid) (day 16 to 22, last dose on morning of day 22)
Arm/Group | Tenofovir | Tenofovir/Faldaprevir | Faldaprevir
Number analyzed (Participants) | 16 | 16 | 0
ng*h/mL | 2700 (26.5) [0.00 to 0.00] | 3290 (19.6) [0.00 to 0.00] |
Statistical Analysis 1: Comparison: Tenofovir vs Tenofovir/Faldaprevir; Test type: Superiority or Other; ANOVA; No formal testing. Investigation of relative bioavailability; Geometric mean ratio = 121.89, 90% CI 2-sided [111.714 to 132.999], Standard Deviation 14.1 — The standard deviation is actually the intra-individual geometric coefficient of variation (gCV)

2. Primary Outcome: Steady-state Pharmacokinetics of Cmax of Tenofovir on Day 7 and on Day 15
Description: Maximum measured concentration of analyte in plasma (Cmax), at steady state.
Time Frame: 144:00, 144:30, 145:00, 145:30, 146:00, 147:00, 148:00, 150:00, 152:00, 156:00, 168:00 hours on day 7 and 168:00, 168:30, 169:00, 169:30, 170:00, 172:00, 174:00, 176:00, 178:00, 180:00. 192:00 hours on day 15
Population: All participants from the pharmacokinetic analysis set (PK set), including all subjects in the treated set who provided evaluable data for at least 1 observation for at least 1 primary PK endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Tenofovir: tenofovir medium dose (300mg) once daily (qd) (day 1 to 7
Arm/Group | Tenofovir | Tenofovir/Faldaprevir | Faldaprevir
Number analyzed (Participants) | 16 | 16 | 0
ng/mL | 300 (27.3) | 284 (16.6) |
Statistical Analysis 1: Comparison: Tenofovir vs Tenofovir/Faldaprevir; Test type: Superiority or Other; ANOVA; No formal testing. Investigation of relative bioavailability; Geometric mean ratio = 94.72, 90% CI 2-sided [85.215 to 105.290], Standard Deviation 17.2 — The standard deviation is actually the intra-individual gCV

3. Primary Outcome: Steady-state Pharmacokinetics of C24hr of Tenofovir on Day 7 and on Day 15
Description: Measured concentration of the analyte in plasma at 24 h (C24hr) after dosing, at steady state.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Tenofovir | Tenofovir/Faldaprevir | Faldaprevir
Number analyzed (Participants) | 16 | 16 | 0
ng/mL | 54.0 (26.7) | 79.4 (21.5) |
Statistical Analysis 1: Comparison: Tenofovir vs Tenofovir/Faldaprevir; Test type: Superiority or Other; ANOVA; No formal testing. Investigation of relative bioavailability; Geometric mean ratio = 147.12, 90% CI [134.482 to 160.943], Standard Deviation 14.6 — The standard deviation is actually the intra-individual gCV

4. Primary Outcome: Steady-state Pharmacokinetics of AUC0-12 of Faldaprevir on Day 15 and on Day 22
Description: Area under the concentration-time curve (AUC) of the analyte in plasma over the time interval 0-12 hours, at steady state.
Time Frame: 168:00, 168:30, 169:00, 169:30, 170:00, 172:00, 174:00, 176:00, 178:00, 180:00, 192:00 hours on day 15 and 144:00, 144:30, 145:00, 145:30, 146:00, 147:00, 148:00, 150:00, 152:00, 156:00 hours on day 22
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Tenofovir | Tenofovir/Faldaprevir | Faldaprevir
Number analyzed (Participants) | 0 | 16 | 14
ng*h/mL |  | 418000 (69.3) | 523000 (101)
Statistical Analysis 1: Comparison: Tenofovir/Faldaprevir vs Faldaprevir; Test type: Superiority or Other; ANOVA; No formal testing. Investigation of relative bioavailability; Geometric mean ratio = 77.88, 90% CI 2-sided [71.24 to 85.15], Standard Deviation 13.4 — The standard deviation is actually the intra-individual gCV

5. Primary Outcome: Steady-state Pharmacokinetics of Cmax of Faldaprevir on Day 15 and Day 22
Description: Maximum measured concentration of analyte in plasma (Cmax), at steady state.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Tenofovir | Tenofovir/Faldaprevir | Faldaprevir
Number analyzed (Participants) | 0 | 16 | 14
ng/mL |  | 41700 (51.4) | 50400 (91.3)
Statistical Analysis 1: Comparison: Tenofovir/Faldaprevir vs Faldaprevir; Test type: Superiority or Other; ANOVA; No formal testing. Investigation of relative bioavailability; Geometric mean ratio = 81.73, 90% CI 2-sided [71.56 to 93.34], Standard Deviation 20.1 — The standard deviation is actually the intra-individual gCV

6. Primary Outcome: Steady-state Pharmacokinetics of C12hr of Faldaprevir on Day 15 and on Day 22
Description: Measured concentration of the analyte in plasma at 12 h (C12hr) after dosing, at steady state.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Tenofovir | Tenofovir/Faldaprevir | Faldaprevir
Number analyzed (Participants) | 0 | 16 | 14
ng/mL |  | 31000 (79.5) | 40000 (113)
Statistical Analysis 1: Comparison: Tenofovir/Faldaprevir vs Faldaprevir; Test type: Superiority or Other; ANOVA; No formal testing. Investigation of relative bioavailability; Geometric mean ratio = 75.27, 90% CI 2-sided [68.71 to 82.45], Standard Deviation 13.7 — The standard deviation is actually the intra-individual gCV

7. Secondary Outcome: Number of Patients With Drug Related Adverse Events During the Trial
Description: Outcome data are the numbers of subjects with investigator defined drug-related AEs
Time Frame: From drug administration up to 32 days.
Population: All subjects who were dispensed study medication and were documented to have taken at least one dose of study drug were included in the safety evaluation (treated set).
Measure: Number; unit: participants
Arm/Group | Tenofovir | Tenofovir/Faldaprevir | Faldaprevir
Number analyzed (Participants) | 16 | 16 | 16
participants | 0 | 15 | 9

8. Secondary Outcome: Clinical Relevant Abnormalities for Physical Examination, Vital Signs, Safety Laboratory Tests and 12-lead ECG
Description: Clinical relevant abnormalities for physical examination, vital signs, safety laboratory tests and 12-lead ECG. New abnormal findings or worsening of baseline conditions were reported as Adverse Events.
  Preferred term of relevant AE: Presyncope
Time Frame: From drug administration up to 32 days.
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Tenofovir | Tenofovir/Faldaprevir | Faldaprevir
Number analyzed (Participants) | 16 | 16 | 16
participants | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From drug administration up to 32 days
Arm/Group | Tenofovir | Tenofovir/Faldaprevir | Faldaprevir
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 16/16 | 10/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir (N=16) | Tenofovir/Faldaprevir (N=16) | Faldaprevir (N=16)
Oral herpes (Infections and infestations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 10 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Ocular icterus (Eye disorders) | 0 | 3 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 7 | 1
Nausea (Gastrointestinal disorders) | 0 | 6 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 2 | 1
Pain (General disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.